CLINICAL TRIAL: NCT05512442
Title: Comparison of the Centric Relation Recorded by the Gothic Arch Methods and the Neuromuscular Method Using Cone Beam Computed Tomography
Brief Title: Comparison of the Centric Relation Recorded by Two Methods Using Cone Beam Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20200901
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Tooth Loss
Keywords: Cone-Beam computed tomography; the centric relation; the upper airway; mandibular position
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- record the centric relation using the gothic tracing method (Experimental): the vertical dimension of occlusion (VDO) were were determineded through facial appearance observation,thus,the patients were trained to execute bordering protrusive, retrusive and bilateral lateral-protrusive movements wearing the intraoral apparatus and a Gothic Arch Tracing was made, the apex of the Gothic Arch Tracing was defined as the gothic arch position.
  Interventions: Procedure: the centric relation
- record the centric relation using the neuromuscular method (Experimental): the participant were subjected to a low-frequency transcutaneous electrical nerve stimulation (TENS) using the J5 Myotronics for 45 minutes,With the help of TENS, complete relaxation of the muscles were achieved and the mandibular musculature was induced to guide the mandible in the physiologic position,thus using K7 to track the physical mandibular positon which was defined as the neuromuscular position.
  Interventions: Procedure: the centric relation

INTERVENTIONS:
Procedure: the centric relation — All participants were recorded the centric relation registrations according to the technique of the gothic tracing method and the neuromuscular method separately.

SUMMARY:
The purpose of this study was to investigate and compare the variation in mandibular relation recorded by the gothic arch methods and the K7 method using cone beam computed tomography (CBCT)

DETAILED DESCRIPTION:
ten asymptomatic participants were selected,the centric relation registrations were separately recorded according to the technique of the gothic arch method and the neuromuscular method,subsequent, they were instructed to perform CBCT wearing two bite registrations,thus using dophin software to calculate the tmj space and the upper airway and using exocad software to ananyse the mandibular position, Data were analysed with paired t-test

ELIGIBILITY:
Inclusion Criteria:

absence of the mandibular position Classified as ASA 1 or 2 (normal healthy patient or with mild systemic disease, according to the American Society of Anaesthesiologists Physical Status Classification System); Absence of the symptoms and signs of the temporomandibular joint; Willing to participate and to sign a written informed consent form.

Exclusion Criteria:

Cardiac pacemaker carriers and pregnant women; people with heart pace disorders and epilepsy; Temporomandibular or craniocervical disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
the temporomandibular joint space | immediately
  according to the method of Ikeda and Kawamura, tmj space measurement in sagittal of the CBCT images were performed

SECONDARY OUTCOMES:
the upper airway | immediately
  Using the sinus/airway feature of the Dolphin software to reconstruct the upper airway,it included three region: the nasopharynx, oropharynx, and hypopharynx

OTHER OUTCOMES:
the mandibular position | immediately
  convert the DICOM files into the exocad software and analyse the difference of the mandibular position determined by the technique of the gothic tracing method and the neuromuscular method separately.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No